CLINICAL TRIAL: NCT02514187
Title: A Blinded Study Evaluating the Accuracy and Safety of Cyclotron-produced 99mTc in Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Centre for Probe Development and Commercialization (Other); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other); TRIUMF (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Natural Resources, Canada (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: H15-01132
Record Dates: First submitted 2015-07-27; First posted 2015-08-03 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2018-12

CONDITIONS: Hyperthyroidism
Keywords: Osteogenesis
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evaluation of hyperthyroidism (Other): For the evaluation of hyperthyroidism each research subject will undergo imaging using both cyclotron-produced 99mTc and the current standard method used at the site for thyroid imaging (either 123I or generator-produced 99mTc). Each study will be performed on a separate day, with flexibility to schedule either study first.
  Interventions: Drug: Cyclotron-produced 99mTc; Drug: Generator-produced 99mTc
- Evaluation of altered osteogenesis by bone scintigraphy (Other): For the evaluation of altered osteogenesis by bone scintigraphy each research subject will serve as his/her own control, and undergo imaging using both generator- and cyclotron-produced 99mTc. Each study will be performed on a separate day, with flexibility to schedule either study first.
  Interventions: Drug: Cyclotron-produced 99mTc; Drug: Generator-produced 99mTc

INTERVENTIONS:
Drug: Cyclotron-produced 99mTc — Each research subject will serve as his/her own control, and will undergo imaging using both generator- and cyclotron-produced 99mTc. The study will follow the usual clinical procedure for routine imaging in the nuclear medicine department.
  All subjects will be contacted by phone or in person the day following the injection of both generator and cyclotron-produced 99mTc to monitor for potential adverse events.
Drug: Generator-produced 99mTc — Each research subject will serve as his/her own control, and will undergo imaging using both generator- and cyclotron-produced 99mTc. The study will follow the usual clinical procedure for routine imaging in the nuclear medicine department.
  All subjects will be contacted by phone or in person the day following the injection of both generator and cyclotron-produced 99mTc to monitor for potential adverse events.

SUMMARY:
The purpose of this study is to evaluate technetium-99m (99mTc) pertechnetate produced by a cyclotron as a replacement for 99mTc pertechnetate obtained from a generator containing the parent isotope Molybdenum-99 (99Mo). 99mTc pertechnetate is currently used in nuclear medicine departments across the country. 99Mo is produced by a number of ageing nuclear reactors across the world and severe shortages of the isotope have occurred in the past few years. Cyclotron-produced 99mTc offers an alternative decentralized production method on a regional basis. Since the manufacturing process is different, the safety and efficacy of cyclotron-produced 99mTc pertechnetate must be evaluated in human subjects to enable its routine clinical use.

ELIGIBILITY:
Inclusion Criteria:

* WHO performance status 0-2
* Older than the age of majority in the province where the study is performed, and be able to consent to the project
* Ambulatory and able to lie supine for the duration of the examination.
* Able and willing to return for a subsequent visit within 7 days to undergo a repeat examination and participate in a follow-up phone call to monitor for adverse events.

Subject referred for nuclear medicine examination for one of the following indications:

* Biochemically documented hyperthyroidism, referred for scintigraphy to evaluate the differential diagnosis of hyperthyroidism or to plan radioiodine treatment.
* Referred for bone scintigraphy for the evaluation of metastases, fractures, or inflammatory conditions. Subjects referred for a limited area (localized) bone scan are eligible, provided they agree to undergo a whole-body scan as part of the procedure.

Exclusion Criteria:

* Pregnant, planning to become pregnant within 30 days
* Severe evolving health problems (unstable coronary disease, liver failure, heart failure, end-stage-renal failure, hospitalized subjects with severe medical conditions) that may confound the assessment of adverse events.

For subjects evaluated for hyperthyroidism:

* Recent iodine-containing IV contrast administration (< 6 weeks)
* Recent amiodarone usage (< 8 weeks)

For subjects evaluated for bone scintigraphy:

• Recent trauma occurring less than 24 hours prior to the first 99mTc bone scintigraphy examination, or between the first and second 99mTc bone scintigraphy examination.

Women who are breast-feeding are eligible to participate in this study, but must cease breast-feeding for 24 hours following the 99mTc examinations. They can draw their milk and discard it during this period, and use either formula or previously collected milk to feed their child.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Agreement rate of the blinded read of scintiscans between cyclotronproduced 99mTc (CP) and the standard of care (SOC) in the diagnosis of hyperthyroidism | 12 weeks
  The result of the standard of care test and cyclotron-produced 99mTc pertechnetate will be compiled in a 2 x 2 table, and the corresponding proportions will be compared.
  The accuracy of the thyroid examinations will be compared to a clinical standard of care consisting of a combination of physical examination, laboratory testing, ultrasound evaluation (when available) and short-term clinical follow-up at 12 weeks. The accuracy of cyclotron-produced 99mTc will be compared to the accuracy of generator-produced 99mTc or 123I, using a non-inferiority test of correlated proportions.

SECONDARY OUTCOMES:
Blinded subjective comparison of image quality between cyclotron- and generator-produced 99mTc using a 5-point Likert scale. | 1 year
  For the subjective evaluation of image quality, data will be scored on a 5-point Likert scale, evaluating independently and blindly cyclotron- and generator-produced 99mTc. The scores on this ordinal scale will be compared using a one-sided Mann-Whitney test for paired samples.
The target-to-background ratio | 1 year
  For quantitative evaluation of image contrast, the target-to-background ratio will be calculated by measuring the activity in the organ of interest (long bones). The target-to-background ratios will be compared using a one-sided paired t-test.
Number of participants with 99mTc-related adverse events as assessed by abnormal vital sign measurement. | 1 hour
  Vital signs (blood pressure, heart rate and pulse oximetry) will be measured at three time points (before and after injection, and 1 hour after the injection). All values that fall outside of the normal parameters will be assessed by a physician and reported as an adverse event.
Number of participants with self-reported 99mTc-related adverse event. | 24 hours
  Patients will be contacted by phone 24 hours after the 68Ga-DOTATOC PET/CT scan to see if they experienced any adverse events. These are recorded and evaluated for severity and likelihood they are related to the study drug. All adverse events will be recorded and summarized in the final report.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Benard, MD, Principal Investigator — BC Cancer
Locations (3):
- Canada (3):
  - Vancouver General Hospital - Nuclear Medicine, Vancouver, British Columbia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - London Regional Health Sciences Centre, London, Ontario